CLINICAL TRIAL: NCT01273922
Title: Phase I Double-Blind, Placebo-Controlled Dose Escalation Study to Evaluate the Safety, Tolerability and Immunogenicity of NDV-3, a Recombinant Alum-Adjuvanted Vaccine for Staphylococcus Aureus and Candida Infections, Administered Intramuscular to Healthy Adults
Brief Title: Safety and Immunogenicity Study of a Recombinant Protein Vaccine (NDV-3) Against S.Aureus and Candida
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NovaDigm Therapeutics, Inc. (Industry)
Collaborators: Cetero Research, San Antonio (Network); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NDV-3-001
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Staphylococcal Infections; Candidiasis
Keywords: NDV-3; vaccine; Staphylococcus aureus; MRSA; Candida
MeSH Terms: conditions — Staphylococcal Infections; Candidiasis; Torulopsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Low Dose NDV-3 investigational vaccine (Placebo Comparator): 15 subjects will receive vaccine and 5 subjects will receive placebo.
  Interventions: Biological: NDV-3 investigational vaccine
- High Dose NDV-3 investigational vaccine (Placebo Comparator): 15 subjects will receive vaccine and 5 subjects will receive placebo
  Interventions: Biological: NDV-3 investigational vaccine

INTERVENTIONS:
Biological: NDV-3 investigational vaccine — Two doses of vaccine 6 months apart or placebo(only one dose at Time 0) administered intramuscularly

SUMMARY:
This randomized, double-blind, placebo-controlled study is a first-in-human Phase 1 study using two dose levels of an investigational vaccine directed against S. aureus and Candida. The study is designed to evaluate the safety, tolerability and immunogenicity of the investigational vaccine, NDV-3

DETAILED DESCRIPTION:
Preclinical studies in mice have established that several members of the Als family of proteins induce a protective immune response in mice and allow high survival rates following challenge with highly virulent doses of either Candida or S. aureus. Als3 (the antigen in the NDV-3 investigational vaccine) is the most effective member of the Als protein family in protecting mice from challenge with either Candida or S. aureus. This Phase I study will evaluate the safety and immunogenicity of a two doses administered 6 months apart of NDV-3 vaccine at two dose levels. At least 40 subjects will be enrolled in the study in two groups of approximately 20 subjects each. Each group will be randomized so that 15 will receive NDV-3 vaccine and 5 will receive placebo. All injections will be administered intramuscularly. One group will receive a low dose of NDV-3 and the other a ten-fold higher dose. Subjects will have follow-up visits to assess the safety, tolerability and immune responses at days 3, 7, 14, 28, 90 and 180 after the first vaccination to compare to baseline levels and at days 7, 14 and 90 after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the nature of the study and have agreed to and are able to read, review, and sign the informed consent document prior to screening. The informed consent document will be written in English, therefore the subject must have the ability to read and communicate in English.
2. Completed the screening process within 30 days prior to dosing.
3. Healthy male and female subjects 18-50 years of age, inclusive, at the time of dosing.
4. No clinically significant deviation from normal as judged by the investigator(s) in the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations.
5. Female subjects must be:

   * of childbearing potential and practicing an acceptable method of birth control described below as judged by the investigator(s); or
   * of postmenopausal status (no menses) for at least 1 year and has a documented FSH level ≥ 40 mIU/mL; or
   * sterile (surgically [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy] or the Essure® Procedure).

Exclusion Criteria:

1. Reports receiving any investigational drug, investigational vaccine, or investigational device within 30 days prior to dosing.
2. Reports any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease as determined by the clinical investigator(s).
3. Clinical laboratory test values outside the accepted range.
4. When confirmed upon additional testing, demonstrates a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
5. Reports a clinically significant illness during the 28 days prior to dosing (as determined by the clinical investigators).
6. Demonstrates a positive drug screen for non-prescription drugs.
7. Reports a history of allergic response(s) to nickel or anaphylaxis (or other serious reactions) to aluminum.
8. Reports receiving any live attenuated vaccine including FluMist® within 6 weeks prior to dosing or any licensed inactivated vaccine within 3 weeks prior to dosing.
9. Reports the use of any immunosuppressive drugs, including systemic corticosteroids, within 4 weeks prior to dosing.
10. Reports the use of any medications or treatments that may alter immune responses to the study vaccine within 3 weeks prior to dosing (e.g., cyclosporine, tacrolimus, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin [BCG], monoclonal antibodies, radiation therapy).
11. Reports a history of clinically significant allergies including food or drug allergies or anaphylaxis (or other serious reactions) to vaccines.
12. Reports a history of drug or alcohol addiction or abuse within the past year.
13. Reports receiving any blood products within 3 months prior to dosing and throughout the study.
14. Reports donating blood within 28 days prior to dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
15. Reports donating plasma (e.g. plasmapheresis) within 14 days prior to dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
16. Reports an intolerance of direct venipuncture.
17. Pregnant, lactating, breastfeeding, or intends to become pregnant over the course of the study (females only).
18. Demonstrates a positive pregnancy screen (females only).
19. Any other medical and/or social (e.g. non-compliant) reason which, in the opinion of the investigator(s), would prevent participation in the study.

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the safety and tolerability of one dose of NDV-3 vaccine compared to placebo at two different dose levels. | 1 month
  Clinical evaluations and safety laboratories

SECONDARY OUTCOMES:
The secondary objective is to compare the humoral and cellular immune responses between the two dose levels compared to placebo at several time points over a 6 month period. | 180 days post-injection
  Immune responses to NDV-3 investigational vaccine up to day 180 compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero, Fargo, North Dakota, United States